CLINICAL TRIAL: NCT02553369
Title: Seroprevalence of Chikungunya at the End of the First Chikungunya Outbreak in the French Antilles Within a Sample of Patients Treated for a HIV Infection
Acronym: ChikVIH
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 14/B/18; 2014-A01504-43 (Registry Identifier: ID RCB); 2014/82 (Registry Identifier: N° CPP)
Record Dates: First submitted 2015-09-14; First posted 2015-09-17 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: HIV Infections; Chikungunya Virus Infection
MeSH Terms: conditions — HIV Infections; Chikungunya Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enrolled patients: Patient randomly enrolled in the study within a cohort of patient followed for HIV infection.
  Interventions: Other: Biological sample collection

INTERVENTIONS:
Other: Biological sample collection — A blood sample is collected during a follow up visit for HIV infection.

SUMMARY:
Late 2013, the first indigenous cases of chikungunya have been observed in the French Antilles. At the end of May 2014, almost all of the islands of the Caribbean were affected by the outbreak.

During the large epidemic which affected the Island of La Réunion in 2005/2006, the attack rate was 38%. The most active period was three months.

In this context, knowledge of the attack rate and the epidemic in the Caribbean is an important issue for outbreak management and modeling work.

As the chikungunya virus had never circulated in the Caribbean, determining the seroconversion rate can be achieved by realizing a seroprevalence survey among the general population at the end of the outbreak. Another simple method is to estimate the rate in a cohort of patients followed regularly and whose habitat is distributed throughout the territory studied.

The follow up of patients infected by the human immunodeficiency virus (HIV) in the French West Indies is almost exclusively performed in hospitals in department of Infectious and Tropical Diseases.The high prevalence of HIV and homogeneous distribution of infected patients on all of our territories, allow to hypothesize that the risk of transmission of arboviruses by exposure to mosquito bites is comparable to the general population. This patient cohort is well suited to study the emergence of Chikungunya in the French West Indie .

Primary objective :

To estimate the cumulative incidence at the end of the first Chikungunya outbreak in the French West Indies by estimating the prevalence of specific antibodies of chikungunya virus in a sample (randomly constituted) from patients infected by HIV and representative of the general population of Martinique and Guadeloupe

Secondary objective :

To estimate the frequency of asymptomatic infections by the chikungunya virus in the studied population To estimate the frequency of chronic forms of chikungunya in the studied population

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years old)
* Followed for HIV infection at the 2 investigators centers (1 located at Martinique and 1 at Guadeloupe)
* resident in Martinique /Guadeloupe ( French West Indies)
* informed consent signed by the patient

Exclusion Criteria:

* patient who lived more than 6 month in an risk area for chikungunya virus infection
* patient with or documented chronic rheumatism
* patient who has received a blood transfusion during year 2013 or patient who is supposed to receive a blood transfusion during the study
* patient who has planned to live outside French West Indies during the follow up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient followed for HIV infection at the 2 investigator centers.
Sampling Method: Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Presence or not of chikungunya virus-specific immunoglobulin G antibodies (Elisa test) | 1 day
  Presence or not of chikungunya virus-specific immunoglobulin G antibodies

SECONDARY OUTCOMES:
Change From Baseline in Pain | 6 , 12 , 18 months after the first symptoms of chikungunya virus infection
  Score range from 0 (No pain) to 10 (worst possible pain)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Guadeloupe, Pointe à Pitre, Guadeloupe
  - Centre Hospitalier Universitaire de Fort-de-France, Fort-de-France, Martinique

REFERENCES:
- [Background] Pialoux G, Gauzere BA, Jaureguiberry S, Strobel M. Chikungunya, an epidemic arbovirosis. Lancet Infect Dis. 2007 May;7(5):319-27. doi: 10.1016/S1473-3099(07)70107-X. PMID 17448935
- [Background] Farnon EC, Sejvar JJ, Staples JE. Severe disease manifestations associated with acute chikungunya virus infection. Crit Care Med. 2008 Sep;36(9):2682-3. doi: 10.1097/CCM.0b013e3181843d94. No abstract available. PMID 18728479
- [Background] Brouard C, Bernillon P, Quatresous I, Pillonel J, Assal A, De Valk H, Desenclos JC; workgroup "Quantitative Estimation of the Risk of Blood Donation Contamination by Infectious Agents". Estimated risk of Chikungunya viremic blood donation during an epidemic on Reunion Island in the Indian Ocean, 2005 to 2007. Transfusion. 2008 Jul;48(7):1333-41. doi: 10.1111/j.1537-2995.2008.01646.x. Epub 2008 Feb 22. PMID 18298600
- [Background] Liumbruno GM, Calteri D, Petropulacos K, Mattivi A, Po C, Macini P, Tomasini I, Zucchelli P, Silvestri AR, Sambri V, Pupella S, Catalano L, Piccinini V, Calizzani G, Grazzini G. The Chikungunya epidemic in Italy and its repercussion on the blood system. Blood Transfus. 2008 Oct;6(4):199-210. doi: 10.2450/2008.0016-08. PMID 19112735
- [Background] Sissoko D, Moendandze A, Malvy D, Giry C, Ezzedine K, Solet JL, Pierre V. Seroprevalence and risk factors of chikungunya virus infection in Mayotte, Indian Ocean, 2005-2006: a population-based survey. PLoS One. 2008 Aug 26;3(8):e3066. doi: 10.1371/journal.pone.0003066. PMID 18725980
- [Background] Appassakij H, Khuntikij P, Kemapunmanus M, Wutthanarungsan R, Silpapojakul K. Viremic profiles in asymptomatic and symptomatic chikungunya fever: a blood transfusion threat? Transfusion. 2013 Oct;53(10 Pt 2):2567-74. doi: 10.1111/j.1537-2995.2012.03960.x. Epub 2012 Nov 26. PMID 23176378
- [Background] Bianco C. Dengue and Chikungunya viruses in blood donations: risks to the blood supply? Transfusion. 2008 Jul;48(7):1279-81. doi: 10.1111/j.1537-2995.2008.01806.x. No abstract available. PMID 18651905
- [Background] Ramful D, Carbonnier M, Pasquet M, Bouhmani B, Ghazouani J, Noormahomed T, Beullier G, Attali T, Samperiz S, Fourmaintraux A, Alessandri JL. Mother-to-child transmission of Chikungunya virus infection. Pediatr Infect Dis J. 2007 Sep;26(9):811-5. doi: 10.1097/INF.0b013e3180616d4f. PMID 17721376
- [Background] Gerardin P, Barau G, Michault A, Bintner M, Randrianaivo H, Choker G, Lenglet Y, Touret Y, Bouveret A, Grivard P, Le Roux K, Blanc S, Schuffenecker I, Couderc T, Arenzana-Seisdedos F, Lecuit M, Robillard PY. Multidisciplinary prospective study of mother-to-child chikungunya virus infections on the island of La Reunion. PLoS Med. 2008 Mar 18;5(3):e60. doi: 10.1371/journal.pmed.0050060. PMID 18351797
- [Background] Gerardin P, Guernier V, Perrau J, Fianu A, Le Roux K, Grivard P, Michault A, de Lamballerie X, Flahault A, Favier F. Estimating Chikungunya prevalence in La Reunion Island outbreak by serosurveys: two methods for two critical times of the epidemic. BMC Infect Dis. 2008 Jul 28;8:99. doi: 10.1186/1471-2334-8-99. PMID 18662384
- [Background] Van Bortel W, Dorleans F, Rosine J, Blateau A, Rousset D, Matheus S, Leparc-Goffart I, Flusin O, Prat C, Cesaire R, Najioullah F, Ardillon V, Balleydier E, Carvalho L, Lemaitre A, Noel H, Servas V, Six C, Zurbaran M, Leon L, Guinard A, van den Kerkhof J, Henry M, Fanoy E, Braks M, Reimerink J, Swaan C, Georges R, Brooks L, Freedman J, Sudre B, Zeller H. Chikungunya outbreak in the Caribbean region, December 2013 to March 2014, and the significance for Europe. Euro Surveill. 2014 Apr 3;19(13):20759. doi: 10.2807/1560-7917.es2014.19.13.20759. No abstract available. PMID 24721539
- [Derived] Curlier E, Fagour L, Herrmann-Storck C, Staelen A, Vingadassalom I, Breurec S, Abel S, Pierre-Francois S, Jean-Marie J, Laouenan C, Cesaire R, Hoen B, Cabie A. Seroprevalence of chikungunya virus infection among HIV-infected adults in French Caribbean Islands of Martinique and Guadeloupe in 2015: A cross-sectional study. PLoS Negl Trop Dis. 2021 Apr 9;15(4):e0009267. doi: 10.1371/journal.pntd.0009267. eCollection 2021 Apr. PMID 33836004